CLINICAL TRIAL: NCT00253435
Title: I-Metaiodobenzylguanidine (MIBG) With Intensive Chemotherapy and Autologous Stem Cell Rescue for High-Risk Neuroblastoma
Brief Title: N2001-02: I-MIBG With Intensive Chemotherapy and Autologous Stem Cell Rescue for High-Risk Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nant Operations Center, NANT Operations Center, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000450148; P01CA081403 (NIH); N2001-02 (Other: NANT Consortium)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Carboplatin; Etoposide; etoposide phosphate; Melphalan; 3-Iodobenzylguanidine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All the patients enrolled in the study (Experimental): This is a single arm study. The following description applies to all the patients who are enrolled in the study:
  On Day -21, patients receive 131I-MIBG infusion.
  On Day -7, Day -6, Day -5, patients receive Carboplatin, Etoposide, Melphalan.
  On Day -4, patients receive Carboplatin, Etoposide.
  On Day -3, Day -2, Day -1, patients rest.
  On Day 0, patients receive peripheral blood stem cell infusion.
  Dosing of Carboplatin, Etoposide and Melphalan is based upon whole body dosimetry (cGy) estimates.
  Filgrastim 5 micrograms/kg/day S.C. or IV will be given daily beginning on Day 0.
  Local radiation therapy is to be given to previously non-irradiated primary and metastatic sites of disease.
  Interventions: Biological: Filgrastim; Drug: Carboplatin; Drug: Etoposide; Drug: Melphalan; Procedure: Peripheral blood stem cell infusion; Radiation: 131I-MIBG; Radiation: Radiation therapy

INTERVENTIONS:
Biological: Filgrastim — Filgrastim 5 micrograms/kg/day S.C. or IV will be given daily beginning on Day 0. The first dose should begin four hours after the stem cell infusion is completed. Filgrastim will continue daily until the ANC >=1500/uL for three consecutive days.
  Other Names: G-CSF
Drug: Carboplatin — The carboplatin will be administered as a continuous IV infusion Day - 7 through Day - 4, with dosing based upon pretreatment GFR levels. The carboplatin should be diluted to a concentration of 0.3 mg/ml in D5W 0.45NS and infused concomitantly with etoposide through the same central venous catheter using a "Y" connector; a controlled rate infusion pump is used for each arm of the "Y".
  Other Names: cis-diammine; Paraplatin; Paraplatin-AQ
Drug: Etoposide — The etoposide shall be administered day -7 through day -4 via continuous intravenous infusion over 96 hours. For patients with a corrected GFR >= 100 ml/min/1.72 m^2, a dose of 300 mg/m^2/day (10 mg/kg/day if child is < 12 kg) shall be given. For patients with a corrected GFR 60-99 ml/min/1.72 m^2, the etoposide will be administered at a dose of 160 mg/m^2/day (5.3 mg/kg/day). The etoposide will be diluted in D5W 0.45%NS at a concentration of < 0.4 mg/ml. Etoposide should not be mixed with carboplatin, but administered using a Y-connector.
  Other Names: VP-16; Etopophos
Drug: Melphalan — For patients in either the normal GFR strata (>=100 ml/min/1.73 m^2), or reduced GFR strata (60-99 ml/min/1.73m^2), melphalan shall be administered at a dose of 60 mg/m^2/day (2 mg/kg/day if child is < 12 kg) on day -7, -6, and -5 of study. The melphalan should be infused at a rate of less than 10 mg/minute, and should complete within 1 hour of reconstitution each day. The melphalan should be diluted in 0.9% NaCl at a concentration < 2 mg/ml. The total dosage of melphalan to be administered will be 180 mg/m^2.
  Other Names: L-phenylalanine mustard; L-PAM; Alkeran; Sarcolysin
Procedure: Peripheral blood stem cell infusion — Stem cells or marrow will be infused on day 0 of study therapy. Where the DMSO concentration in the stem cell product would exceed accepted level for infusion within a 24 hour period, stem cell products may be infused over two days to meet this standard. For purged PBSC: A minimum of 2.0 x 10^6 viable CD34+ cells/kg must be available. For unpurged PBSC, a minimum of 2.0 x 10^6 viable CD34+ cells/kg must be available. Having a back-up of 2.0 x 10^6 viable CD34+ cells/kg purged or unpurged PBSC is recommended but not required. For purged bone marrow, a minimum of 1.5 x10^8 mononuclear cells/kg must be available.
Radiation: 131I-MIBG — Therapeutic 131I MIBG will be synthesized by Draximage Canada.with specific activity between 15 and 25mCi/ml. Radiopurity will be initially determined by Draximage, prior to shipment to participating centers. Free radioiodide content must then be rechecked at the treating center prior to infusion using HPLC or Sep-Pac methodology.
  Other Names: Iobenguane I 131
Radiation: Radiation therapy — Local irradiation is to be given to previously non-irradiated primary and metastatic sites of disease. Local irradiation should not start till the patient is medically stable, has an ANC > 1000/uL, platelets > 30,000 / uL, and is > 42 days post transplant. Recommended radiation guidelines consist of 2160 cGy total, given over 12 days using a single 180 cGy fraction/day. Any delay in local radiation that would extend treatment beyond day +84 should be discussed with the study chair. Local radiation will be administered at a participating NANT member site.

SUMMARY:
RATIONALE: Radioactive drugs, such as iodine I 131 metaiodobenzylguanidine, may carry radiation directly to tumor cells and not harm normal cells. Drugs used in chemotherapy, such as carboplatin, etoposide, and melphalan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. An autologous peripheral stem cell or bone marrow transplant may be able to replace blood-forming cells that were destroyed by chemotherapy and radiation therapy. Giving iodine I 131 metaiodobenzylguanidine and combination chemotherapy with an autologous peripheral stem cell or bone marrow transplant may allow more chemotherapy to be given so that more tumor cells are killed. Giving radiation therapy after an autologous peripheral stem cell or bone marrow transplant may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well giving iodine I 131 metaiodobenzylguanidine together with combination chemotherapy and radiation therapy works in treating patients who are undergoing an autologous peripheral stem cell or bone marrow transplant for relapsed or refractory neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with relapsed or refractory neuroblastoma treated with iodine I 131 metaiodobenzylguanidine (^131I-MIBG) and combination chemotherapy comprising carboplatin, etoposide, and melphalan followed by autologous bone marrow or peripheral blood stem cell transplantation and radiotherapy.

Secondary

* Determine the hematopoietic and nonhematopoietic toxicity of this regimen in these patients.
* Determine the tumor self-absorbed radiation dose (TSARD) in patients with measurable soft tissue lesions treated with this regimen.
* Correlate the TSARD with tumor response in patients with measurable residual soft tissue disease treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to risk (poor-risk group [mixed or no response to induction therapy or progression during or after induction therapy] vs good-risk group [partial response after 4 courses of induction therapy]) and kidney function at study entry (glomerular filtration rate [GFR] ≥ 100 mL/min vs GFR 60-99 mL/min)

* Stem cell harvest: Patients undergo a peripheral blood stem cell harvest or bone marrow harvest provided they have an adequate number of cells available. At least 2 weeks later, patients proceed to iodine I 131 metaiodobenzylguanidine (^131I-MIBG) and combination chemotherapy.
* 131I-MIBG and combination chemotherapy: Patients receive ^131I-MIBG IV over 2 hours on day -21, carboplatin IV continuously on days -7 to -4, etoposide IV continuously on days -7 to -4, and melphalan IV over 1 hour on days -7 to -5.
* Stem cell infusion and filgrastim (G-CSF): Three days after completion of chemotherapy, patients undergo transplantation of either stem cells or bone marrow on day 0. Patients also receive G-CSF subcutaneously or IV over 1 hour once daily beginning on day 0 and continuing until blood counts return to normal.
* Radiotherapy: Once blood counts return to normal, patients undergo radiotherapy to primary and metastatic sites that have not received previous irradiation over 12 days beginning after day 42.

After completion of study treatment, patients are followed for 2 years and then periodically thereafter.

PROJECTED ACCRUAL: Approximately 50 patients (40 low-risk patients and 8-10 high-risk patients) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of relapsed or refractory neuroblastoma

  * Histologically confirmed and/or demonstration of tumor cells in bone marrow with elevated urinary catecholamine metabolites
  * High-risk neuroblastoma must meet one of the following:

    * Progressive disease prior to or after completion of induction therapy
    * Mixed response or no response after completion of 4 courses of induction therapy
    * Partial response after 4 courses of induction therapy allowed provided no prior participation in COG-A3973 or other phase III COG trials
* Measurable disease, defined as at least one metaiodobenzylguanidine (MIBG)-avid target lesion determined by diagnostic MIBG scan within 6 weeks of study entry (tumor sites that have received local irradiation within 3 months of study entry are not considered target lesions)

PATIENT CHARACTERISTICS:

Performance status

* Lansky 60-100% OR
* Karnofsky 60-100%

Life expectancy

* At least 2 months

Hematopoietic

* Hemoglobin ≥ 10 g/dL
* Absolute neutrophil count ≥ 750/mm^3
* Platelet count ≥ 50,000/mm^3 (if no marrow involvement by morphologic exam/no transfusion allowed) (> 20,000/mm^3 if metastatic tumor involvement of marrow by morphologic exam/transfusion allowed)

Hepatic

* Bilirubin < 1.3 mg/dL
* SGOT and SGPT < 5 times normal
* Hepatitis B surface antigen negative
* Hepatitis C negative

Renal

* Glomerular filtration rate or creatinine clearance ≥ 60 ml/min
* Creatinine ≤ 1.5 times normal for age as follows:

  * 0.8 mg/dL (for patients ≤ 5 years of age)
  * 1.0 mg/dL (for patients 6 to 10 years of age)
  * 1.2 mg/dL (for patients 11 to 15 years of age)
  * 1.5 mg/dL (for patients > 15 years of age)

Cardiovascular

* Ejection fraction ≥ 55% by echocardiogram or radionuclide MUGA OR
* Fractional shortening ≥ 27% by echocardiogram

Pulmonary

* Normal lung function defined as no dyspnea at rest and no oxygen requirement OR measured oxygen saturation > 93% on room air

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No disease of any major organ system that would preclude study compliance
* No concurrent hemodialysis
* No active infection requiring IV antivirals, antibiotics, or antifungals (patients on antifungal therapy are eligible provided they are culture- and biopsy-negative in suspected residual radiographic lesions)
* Patient weight within limits to receive ≤ maximum total allowable dose of ^131I-MIBG

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior myeloablative transplantation

  * Prior submyeloablative transplantation allowed at discretion of principal investigator
* More than 3 weeks since prior biologic therapy

Chemotherapy

* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for mitomycin C or nitrosoureas)
* No prior melphalan therapy with a total dose of > 100 mg/m^2

Radiotherapy

* See Disease Characteristics
* At least 6 weeks since prior radiotherapy (6 months for craniospinal or whole lung radiotherapy)
* No prior total body irradiation
* No prior iodine I 131 MIBG (^131I-MIBG)
* No prior total abdominal or whole liver radiotherapy
* No prior local radiotherapy, including any of the following:

  * 1200 cGy to more than 33% of both kidneys (patient must have at least one kidney that has not exceeded the dose/volume of radiation listed)
  * 1800 cGy to more than 30% of liver and/or 900 cGy to more than 50% of liver

Other

* Recovered from all prior therapy
* No medications with a potential interference of ^131I-MIBG uptake 1 week before and 2 weeks after completion of ^131I-MIBG

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2005-09; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Yanik, MD, Study Chair — University of Michigan Rogel Cancer Center; Katherine K. Matthay, MD, Principal Investigator — University of California, San Francisco; John M. Maris, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (15):
- United States (14):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Morgan Stanley Children's Hospital of New York-Presbyterian, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Opened to accrual on 12/10/04 & closed to accrual on 07/21/10; suspended 6 times for amendments. Opened at 12 NANT institutions.
  1st patient started on treatment on 03/11/05. 50 patients enrolled; all eligible & evaluable for toxicity. 49 patients were evaluable for response.
Groups:
- Poor Risk Patients: Poor risk patients are those who experienced a Minor response (MR) or No Response (NR) to induction therapy or progressive disease (PD) during or following induction.
- Good Risk Patients: Good risk patients are those who experienced a Partial Response (PR) following 4 cycles of induction.
Period: Overall Study
Arm/Group | Poor Risk Patients | Good Risk Patients
Started | 42 (Total number is 42) | 8 (This cohort opened as long as the poor risk group is open to accrual.)
1st Interim Analysis | 15 (First interim analysis: need 2+ responses in first 15 patients. Goal met study continued.) | 8 (Only interim analysis: need 1+ response in first 10 patients.)
2nd Interim Analysis | 10 (Second interim analysis: need 3+ responses in first 25 patients. Goal met study continued.) | 0 (This cohort opened as long as the poor risk group is open to accrual.)
3rd Interim Analysis | 10 (Third interim analysis: need 4+ responses in first 35 patients. Goal met study continued.) | 0 (This cohort opened as long as the poor risk group is open to accrual.)
Completed | 42 (Forty-two evaluable poor risk patients enrolled.) | 8 (Eight evaluable patients enrolled.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of patients who signed the consent form and started treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Poor Risk Patients | Good Risk Patients | Total
Number analyzed (Participants) | 42 | 8 | 50
Age, Continuous [Median (Full Range); unit: years] — Age (in years) at time of treatment start.
  years | 6.0 [1.1 to 22.8] | 7.7 [4.3 to 16.4] | 6.0 [1.1 to 22.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 32 | 6 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 38 | 5 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 33 | 8 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
GFR Status [Number; unit: participants] — Pre-therapy glomerular filtration rate:
  Normal GFR: >= 100 ml/min/1.73 m2 & Low GFR: 60-99 ml/min/1.73 m2
  participants
    Normal GFR | 30 | 7 | 37
    Low GFR | 12 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Response (Complete Response, Very Good Partial Response, and Partial Response) at 60-days Post Stem Cell Infusion
Description: Tumor response based on evaluation performed on day 60 or at the time of disease progression/recurrence or start of another treatment - whichever comes first. Such evaluations will include 123I-MIBG scan, CT/MRI, urine catecholamine measurement, and bone marrow analysis (for those with marrow disease at study entry).
Time Frame: Response assessed 60 days post stem cell infusion
Population: One patient in the Poor Risk Cohort underwent surgery for resection (of his only measureable lesion) prior to post-treatment assessment and is not evaluable for response.
Measure: Number; unit: participants
Arm/Group | Poor Risk Patients | Good Risk Patients
Number analyzed (Participants) | 41 | 8
participants | 4 | 3

2. Secondary Outcome: Event-free Survival (EFS) at 3 Years
Description: EFS will be measured from start of treatment until progression, death or start of another treatment - whichever comes first. We report the estimated probability of EFS at 3 years.
Time Frame: 3 years since start of treatment
Population: Estimated probability of 3-year progression free survival for all patients enrolled in each risk group.
Measure: Number; unit: Estimated probability
Arm/Group | Poor Risk Patients | Good Risk Patients
Number analyzed (Participants) | 42 | 8
Estimated probability | 0.20 | 0.38

3. Secondary Outcome: Engraftment DLT
Description: • Engraftment toxicity: delayed engraftment and/or failure to engraft defined as:
  * neutrophils (ANC) < 500/μL by day 28 post transplant, or
  * platelets < 20,000 /μL by day 56 post transplant, or
  * if additional stem cells are required to be infused for any medical reason prior to initial engraftment of neutrophils or platelets.
Time Frame: From treatment start until 60 days post stem cell infusion
Population: All patients who began treatment
Measure: Number; unit: participants
Arm/Group | Poor Risk Patients | Good Risk Patients
Number analyzed (Participants) | 42 | 8
participants | 2 | 1

4. Secondary Outcome: Dose Limiting Veno-occlusive Disease (VOD) / Sinusoidal Obstruction Syndrome SOS
Description: Dose limiting veno-occlusive disease (VOD) defined as:
  * the presence of hepatomegaly with right upper quadrant tenderness and an elevation of total bilirubin > grade 1, PLUS
  * the presence of grade 3 abnormalities of any ONE of the following: total bilirubin, hypoalbuminemia, weight gain, or hypoxia without other attribution
Time Frame: Between start of MIBG treatment and 60 days post stem cell infusion
Population: All patients who began treatment
Measure: Number; unit: participants
Arm/Group | Poor Risk Patients | Good Risk Patients
Number analyzed (Participants) | 42 | 8
participants | 6 | 0

ADVERSE EVENTS:
Arm/Group | Poor Risk Patients | Good Risk Patients
Serious Adverse Events (participants affected / at risk) | 12/42 | 3/8
Other Adverse Events (participants affected / at risk) | 42/42 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poor Risk Patients (N=42) | Good Risk Patients (N=8)
Blood/Bone Marrow - Other (DELAYED PLATELET ENGRAFTMENT) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood/Bone Marrow - Other (INFUSION OF BACKUP STEM CELLS) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (2) | 0 (0)
Hepatobiliary/Pancreas - Other (HEPATOMEGALY) (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils (Blood) (Infections and infestations) | 2 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils (Catheter-related) (Infections and infestations) | 1 (1) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 5 (5) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 (0) | 1 (1)
Platelets (Investigations) | 1 (1) | 1 (1)
Weight gain (Investigations) | 5 (5) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Pain (Head/headache) (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poor Risk Patients (N=42) | Good Risk Patients (N=8)
Blood/Bone Marrow - Other (DELAYED ENGRAFTMENT ANC) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Blood/Bone Marrow - Other (INFUSION OF BACKUP SC FOR DELAYED ENGRAFTMENT) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Febrile neutropenia (fever of unknown origin) (Blood and lymphatic system disorders) | 31 (31) | 6 (6) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemoglobin (Blood and lymphatic system disorders) | 40 (40) | 7 (7) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Lymphatics - Other (CAPILLARY LEAK) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Lymphatics - Other (GENERALIZED EDEMA) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Cardiac Arrhythmia - Other (MURMUR) (Cardiac disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Cardiac Arrhythmia - Other (SINUS TACHYCARDIA) (Cardiac disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Cardiac General - Other (SYSTOLIC MURMUR) (Cardiac disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Supraventricular and nodal arrhythmia (Atrial tachycardia/Paroxysmal Atrial Tachycardia) (Cardiac disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Supraventricular and nodal arrhythmia (Sinus tachycardia) (Cardiac disorders) | 11 (11) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Ventricular arrhythmia (Ventricular arrhythmia NOS) (Cardiac disorders) | 0 (0) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (1) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Middle ear) (Ear and labyrinth disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Endocrine - Other (TSH) (Endocrine disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Ocular/Visual - Other (BILATERAL CONJUNCTIVAL HEMORRHAGE) (Eye disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Eye) (Eye disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Ascites (non-malignant) (Gastrointestinal disorders) | 5 (5) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Cheilitis (Gastrointestinal disorders) | 4 (4) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Constipation (Gastrointestinal disorders) | 8 (8) | 2 (2) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dental: teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Diarrhea (Gastrointestinal disorders) | 32 (32) | 4 (4) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Distension/bloating, abdominal (Gastrointestinal disorders) | 5 (5) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Gastrointestinal - Other (HICCUPS) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Gastrointestinal - Other (LOOSE TEETH) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Gastrointestinal - Other (REFLUX) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage, GI (Lower GI NOS) (Gastrointestinal disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage, GI (Oral cavity) (Gastrointestinal disorders) | 2 (2) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage, GI (Stomach) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage, GI (Upper GI NOS) (Gastrointestinal disorders) | 5 (5) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucositis/stomatitis (clinical exam) (Anus) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucositis/stomatitis (clinical exam) (Esophagus) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucositis/stomatitis (clinical exam) (Oral cavity) (Gastrointestinal disorders) | 29 (29) | 5 (5) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucositis/stomatitis (clinical exam) (Rectum) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucositis/stomatitis (functional/symptomatic) (Large bowel) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucositis/stomatitis (functional/symptomatic) (Oral cavity) (Gastrointestinal disorders) | 14 (14) | 4 (4) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucositis/stomatitis (functional/symptomatic) (Small bowel) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucositis/stomatitis (functional/symptomatic) (Stomach) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Nausea (Gastrointestinal disorders) | 32 (32) | 5 (5) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Obstruction, GI (Small bowel NOS) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Abdomen NOS) (Gastrointestinal disorders) | 20 (20) | 3 (3) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Esophagus) (Gastrointestinal disorders) | 1 (1) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Oral cavity) (Gastrointestinal disorders) | 19 (19) | 3 (3) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Oral-gums) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Rectum) (Gastrointestinal disorders) | 1 (1) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Stomach) (Gastrointestinal disorders) | 2 (2) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Salivary gland changes/saliva (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Vomiting (Gastrointestinal disorders) | 33 (33) | 7 (7) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Constitutional Symptoms - Other (BRITTLE HAIR) (General disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Constitutional Symptoms - Other (RHINORRHEA) (General disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Edema:head and neck (General disorders) | 5 (5) | 2 (2) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Edema:limb (General disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Edema:trunk/genital (General disorders) | 2 (2) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Fatigue (asthenia, lethargy, malaise) (General disorders) | 12 (12) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 16 (16) | 2 (2) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Irritability (children <3 years of age) (General disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Chest/thorax NOS) (General disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Face) (General disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Pain NOS) (General disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain - Other (BROVIAC SITE) (General disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain - Other (CVC SITE) (General disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain - Other (GENERAL (NOS)) (General disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain - Other (MOUTH PAIN) (General disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain - Other (MUCOSITIS) (General disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain - Other (OROPHANRIX) (General disorders) | 0 (0) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain - Other (PAROTID GLAND) (General disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain - Other (WHOLE BODY) (General disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Rigors/chills (General disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hepatobiliary/Pancreas - Other (CHOLANGITIS) (Hepatobiliary disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Liver) (Hepatobiliary disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Portal vein flow (Hepatobiliary disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Blood) (Infections and infestations) | 5 (5) | 2 (2) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Catheter-related) (Infections and infestations) | 2 (2) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Lung (pneumonia)) (Infections and infestations) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Mucosa) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Sinus) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Skin (cellulitis)) (Infections and infestations) | 1 (1) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection - Other (ASPERGILLUS OF MOUTH) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection - Other (L-PRESEPTAL CELLULITIS) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection - Other (ORAL CANDIDA) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection - Other (PERIRECTAL CELLULITIS) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection - Other (URINE + FOR CYTOMEGALOVIRUS) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection - Other (VARICELLA) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with normal ANC or Grade 1 or 2 neutrophils (Blood) (Infections and infestations) | 6 (6) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with normal ANC or Grade 1 or 2 neutrophils (Bronchus) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with normal ANC or Grade 1 or 2 neutrophils (Catheter-related) (Infections and infestations) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with normal ANC or Grade 1 or 2 neutrophils (Colon) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with normal ANC or Grade 1 or 2 neutrophils (Lung (pneumonia)) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with normal ANC or Grade 1 or 2 neutrophils (Oral cavity-gums (gingivitis)) (Infections and infestations) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with normal ANC or Grade 1 or 2 neutrophils (Sinus) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with normal ANC or Grade 1 or 2 neutrophils (Small bowel NOS) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with normal ANC or Grade 1 or 2 neutrophils (Upper airway NOS) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with unknown ANC (Catheter-related) (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infection with unknown ANC (Skin (cellulitis)) (Infections and infestations) | 0 (0) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Rash: dermatitis associated with radiation (Chemoradiation) (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 34 (34) | 8 (8) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 36 (36) | 8 (8) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Alkaline phosphatase (Investigations) | 8 (8) | 2 (2) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Bilirubin (hyperbilirubinemia) (Investigations) | 10 (10) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Creatinine (Investigations) | 7 (7) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Fibrinogen (Investigations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 15 (15) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
INR (International Normalized Ratio of prothrombin time) (Investigations) | 7 (7) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Leukocytes (total WBC) (Investigations) | 38 (38) | 8 (8) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Lymphopenia (Investigations) | 30 (30) | 5 (5) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Metabolic/Laboratory - Other (CHLORIDE) (Investigations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Metabolic/Laboratory - Other (DECREASED TOTAL PROTEIN) (Investigations) | 0 (0) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Metabolic/Laboratory - Other (HYPERCHLOREMIA) (Investigations) | 0 (0) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Metabolic/Laboratory - Other (HYPERCHLORIDEMIA) (Investigations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Metabolic/Laboratory - Other (HYPERPHOSPHATEMIA) (Investigations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Metabolic/Laboratory - Other (INCREASED CHLORIDE) (Investigations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Metabolic/Laboratory - Other (INCREASED FIBRINOGEN) (Investigations) | 0 (0) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Metabolic/Laboratory - Other (PRE-ALBUMIN) (Investigations) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 39 (39) | 7 (7) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
PTT (Partial Thromboplastin Time) (Investigations) | 8 (8) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Platelets (Investigations) | 40 (40) | 7 (7) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Weight gain (Investigations) | 10 (10) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Weight loss (Investigations) | 8 (8) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 38 (38) | 8 (8) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Anorexia (Metabolism and nutrition disorders) | 25 (25) | 6 (6) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 8 (8) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 8 (8) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 29 (29) | 6 (6) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 30 (30) | 8 (8) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 16 (16) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 12 (12) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 22 (22) | 6 (6) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 26 (26) | 5 (5) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 12 (12) | 2 (2) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 32 (32) | 7 (7) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 9 (9) | 3 (3) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 34 (34) | 8 (8) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 28 (28) | 6 (6) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Muscle weakness, generalized or specific area (not due to neuropathy) (Extremity-lower) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Muscle weakness, generalized or specific area (not due to neuropathy) (Extremity-upper) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Musculoskeletal/Soft Tissue - Other (NOT SPECIFIED) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Musculoskeletal/Soft Tissue - Other (OCCASIONAL ACHES AND PAINS) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Back) (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Bone) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Chest wall) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Extremity-limb) (Musculoskeletal and connective tissue disorders) | 9 (9) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Joint) (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Neck) (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Neurology - Other (ACHY FEELING) (Nervous system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Neurology - Other (DYSTONIC REACTION) (Nervous system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Neurology - Other (GENERALIZED TENDERNESS) (Nervous system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Neuropathy: cranial (CN VII Motor-face; Sensory-taste) (Nervous system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Neuropathy: motor (Nervous system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Head/headache) (Nervous system disorders) | 5 (5) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Syncope (fainting) (Nervous system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Taste alteration (dysgeusia) (Nervous system disorders) | 4 (4) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Tremor (Nervous system disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Confusion (Psychiatric disorders) | 2 (2) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mood alteration (Agitation) (Psychiatric disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mood alteration (Anxiety) (Psychiatric disorders) | 4 (4) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mood alteration (Depression) (Psychiatric disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 2 (2) | 2 (2) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Bladder spasms (Renal and urinary disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Cystitis (Renal and urinary disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemoglobinuria (Renal and urinary disorders) | 1 (1) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage, GU (Bladder) (Renal and urinary disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage, GU (Urinary NOS) (Renal and urinary disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Bladder) (Renal and urinary disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Proteinuria (Renal and urinary disorders) | 12 (12) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Renal/Genitourinary - Other (DECREASED URINE OUTPUT) (Renal and urinary disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Renal/Genitourinary - Other (FLUID RETENTION) (Renal and urinary disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Pelvis) (Reproductive system and breast disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Penis) (Reproductive system and breast disorders) | 1 (1) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Scrotum) (Reproductive system and breast disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Vaginal mucositis (Reproductive system and breast disorders) | 0 (0) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 2 (2) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage, pulmonary/upper respiratory (Nose) (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage, pulmonary/upper respiratory (Respiratory tract NOS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucositis/stomatitis (clinical exam) (Larynx) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucositis/stomatitis (clinical exam) (Pharynx) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucositis/stomatitis (functional/symptomatic) (Pharynx) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Larynx) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (Throat/pharynx/larynx) (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pulmonary/Upper Respiratory - Other (CONGESTION) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pulmonary/Upper Respiratory - Other (HYPERCARBIA) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pulmonary/Upper Respiratory - Other (RHINORRHEA) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pulmonary/Upper Respiratory - Other (RUNNY NOSE) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pulmonary/Upper Respiratory - Other (TACHYPNEIC) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dermatology/Skin - Other (DRY LIPS) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dermatology/Skin - Other (FACIAL ABRAISIONS) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dermatology/Skin - Other (INGROWN TOENAIL) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dermatology/Skin - Other (LACERATION) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dermatology/Skin - Other (PEELING SKIN) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dermatology/Skin - Other (PERIORBITAL ECCHYMOSES) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dermatology/Skin - Other (PSEUDOMEMBRANOUS CHANGES) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dermatology/Skin - Other (SORE/SCAB) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dermatology/Skin - Other (SUN BURN) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dermatology/Skin - Other (ZOSTER LESION) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pruritus/itching (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Rash/desquamation (Skin and subcutaneous tissue disorders) | 19 (19) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Flushing (Vascular disorders) | 3 (3) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hematoma (Vascular disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage/Bleeding - Other (EPISTAXIS) (Vascular disorders) | 2 (2) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage/Bleeding - Other (EYE) (Vascular disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage/Bleeding - Other (HEMATURIA) (Vascular disorders) | 1 (1) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage/Bleeding - Other (HEMOPTYSIS) (Vascular disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage/Bleeding - Other (NOSE BLEED) (Vascular disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemorrhage/Bleeding - Other (TONGUE BLEED) (Vascular disorders) | 1 (1) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypertension (Vascular disorders) | 8 (8) | 0 (0) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypotension (Vascular disorders) | 13 (13) | 1 (1) — We are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other